CLINICAL TRIAL: NCT00516360
Title: Chlorhexidine and the Prevention of Central Catheter Related Infections in Neonates
Brief Title: Study of Chlorhexidine as the Hub Antiseptic to Prevent Catheter Related Infections in Newborn Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Rochester (Other)
Responsible Party: Erik Thingvoll, MD, University of Rochester Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: T32AI007464 (NIH); 00016854
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2007-08

CONDITIONS: Catheterization
Keywords: Catheter related bloodstream infections; Infant, Newborn; Intensive Care Units, Neonatal; Neonatal Central Line Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Chlorhexidien as the antibacterial agent used to cleanse the hub of neonatal central lines
  Interventions: Device: 3.15% chlorhexidine as daily antiseptic on needleless access port
- 2 (Active Comparator): Isopropyl alcohol as the antibacterial agent used to cleanse the hub of neonatal central lines
  Interventions: Device: 3.15% chlorhexidine as daily antiseptic on needleless access port

INTERVENTIONS:
Device: 3.15% chlorhexidine as daily antiseptic on needleless access port — 3.15% chlorhexidine as daily antiseptic on needleless access port. 1 wipe used to cleanse port each time the port is accessed
  Other Names: Chloraprep

SUMMARY:
The purpose of this study is to prevent catheter-related infections in newborn infants admitted to the Neonatal Intensive Care Unit (NICU). This study will compare the effectiveness of daily chlorhexidine versus isopropyl alcohol in preventing the growth of microbes in catheters.

DETAILED DESCRIPTION:
Catheter-related bloodstream infections (CRBSIs) are a major cause of morbidity and mortality in infants admitted to the NICU. In adults, chlorhexidine used as a skin antiseptic has been shown to reduce the incidence of CRBSIs, and recent evidence indicates the inner surface of long-term central catheters as the likely route of infection. This study will evaluate 3.15% chlorhexidine as the daily catheter hub antiseptic to reduce catheter tip microbial colonization, an indication of high risk for acquiring CRBSI. The purpose of this study is to compare the antiseptic capability of 3.15% chlorhexidine versus isopropyl alcohol in reducing central catheter-related infections in neonates. This study also aims to compare the time to catheter hub microbial colonization in the two groups and to determine the route of catheter tip colonization by comparing cultures taken from the catheter tip, hub, and skin insertion site.

This study will last 1 year. There are no study visits. The placement and removal of the catheter will be determined by the discretion of the attendant caring for the participant. Participants will be randomly assigned to one of two groups. Catheters of Group 1 participants will be treated with 3.15% chlorhexidine at the time of the daily intravenous tubing change. Catheters of Group 2 participants will be treated with isopropyl alcohol. For both groups, cultures of the inner surface of the catheter hub will be performed twice a week, and cultures of the inner surface of the catheter hub, tip, and skin insertion site will be performed upon removal of the catheter.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the NICU
* Umbilical vein catheter or peripherally inserted central venous catheter (PICC) anticipated to be in place for more than 48 hours
* Parent or guardian able to give informed consent prior to first hyperalimentation and total parenteral nutrition tubing change

Exclusion Criteria:

* Known CRBSI-positive blood culture at the time of catheter line placement.
* Not expected to survive for more than 48 hours
* Broviac or any other surgically-placed central catheters
* Any condition that, as determined by the investigator, would interfere with evaluation of the line or be a potential health risk to the participant

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Catheter tip microbial colonization | at the time of catheter removal

SECONDARY OUTCOMES:
Time to hub microbial colonization | at the time of catheter removal
Route of catheter tip microbial colonization determined by cultures taken at the catheter hub versus skin | at the time of catheter removal

CONTACTS AND LOCATIONS:
Overall Officials: Erik S. Thingvoll, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Garland JS, Alex CP, Mueller CD, Otten D, Shivpuri C, Harris MC, Naples M, Pellegrini J, Buck RK, McAuliffe TL, Goldmann DA, Maki DG. A randomized trial comparing povidone-iodine to a chlorhexidine gluconate-impregnated dressing for prevention of central venous catheter infections in neonates. Pediatrics. 2001 Jun;107(6):1431-6. doi: 10.1542/peds.107.6.1431. PMID 11389271
- [Background] Garland JS, Henrickson K, Maki DG; 2002 Hospital Infection Control Practices Advisory Committee Centers for Disease Control and Prevention. The 2002 Hospital Infection Control Practices Advisory Committee Centers for Disease Control and Prevention guideline for prevention of intravascular device-related infection. Pediatrics. 2002 Nov;110(5):1009-13. doi: 10.1542/peds.110.5.1009. No abstract available. PMID 12415044